CLINICAL TRIAL: NCT00823680
Title: Multi-center, Randomized, Double-blind, 5-arm Parallel Group, Placebo Controlled 4 Week Study to Investigate the Safety, Tolerability and Efficacy of Two Doses Each (Near to Maximum Tolerated Dose and Lower Dose) of RO5093151 Administered Twice Daily (BID Regimen) and RO5027838 Administered Once da
Brief Title: A Study of RO5093151 and RO5027838 in Patients With Type 2 Diabetes Mellitus on a Stable Dose of Metformin
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BP21850; 2008-001122-13
Record Dates: First submitted 2009-01-15; First posted 2009-01-16 (Estimated); Last update posted 2016-07-28 (Estimated); Status verified 2016-07

CONDITIONS: Diabetes Mellitus Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (5):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- RO5027838 200mg (Experimental)
  Interventions: Drug: RO5027838
- RO5027838 50mg (Experimental)
  Interventions: Drug: RO5027838
- RO5093151 10mg (Experimental)
  Interventions: Drug: RO5093151
- RO5093151 400mg (Experimental)
  Interventions: Drug: RO5093151

INTERVENTIONS:
Drug: Placebo — po bid for 4 weeks
  Arms: Placebo
Drug: RO5027838 — 200mg po qd for 4 weeks
  Arms: RO5027838 200mg
Drug: RO5027838 — 50mg po bid for 4 weeks
  Arms: RO5027838 50mg
Drug: RO5093151 — 400mg po bid for 4 weeks
  Arms: RO5093151 400mg
Drug: RO5093151 — 10mg po bid for 4 weeks
  Arms: RO5093151 10mg

SUMMARY:
This 5 arm study will evaluate the efficacy and safety of RO5093151 and RO5027838 in patients with type 2 diabetes mellitus on a stable dose of metformin. After a 4 week pre-randomization period for glucose control, patients will be randomized to one of 5 groups to receive a)RO5093151 400mg po bid b)RO5093151 10mg po bid c)RO5027838 200mg po qd d)RO5027838 50mg po qd or e)placebo po bid for 4 weeks. The anticipated time on study treatment is < 3 months, and the target sample size is 100-500 individuals.

ELIGIBILITY:
Inclusion Criteria:

* adult patients, 35-65 years of age;
* type 2 diabetes for >=3 months;
* treated for >=3 months with stable dose of metformin >=1.5g/day or maximum tolerated dose.

Exclusion Criteria:

* history of diabetic ketoacidosis;
* currently or previously treated with insulin;
* currently or within previous 6 months treated with a thiazolidinedione or dual peroxisome proliferator activated receptor (PPAR) agonist;
* treated with lipoprotein-modifying therapy within a month before screening.

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2009-04; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Absolute change in mean daily plasma glucose | From baseline to day 27

SECONDARY OUTCOMES:
Fasting plasma glucose | Baseline, and weeks 1, 2, 3 and 4
Post-prandial glucose and insulin | Baseline, weeks 2 and 4
Insulin sensitivity, beta cell function, lipid profile, HbA1C | At baseline, and at planned visits up to week 4
Adverse events, lab parameters, vital signs, body weight | At baseline, and at planned visits up to week 4

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (5):
- United States (2):
  - Chula Vista, California
  - Miami, Florida
- Graz, Austria
- Germany (2):
  - München
  - Neuss